CLINICAL TRIAL: NCT06932107
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center Phase III Study to Evaluate the Efficacy and Safety of Aprepitant Injection(QLG2174) in the Prevention of Post-operative Nausea and Vomiting
Brief Title: Efficacy and Safety Study of Aprepitant Injection for Prevention of Post-operative Nausea and Vomiting
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical (Hainan) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: QLG2174-301
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Aprepitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aprepitant Injection (Experimental)
  Interventions: Drug: Aprepitant Injection
- Aprepitant Injection Placebo (Experimental)
  Interventions: Drug: Aprepitant Injection Placebo

INTERVENTIONS:
Drug: Aprepitant Injection — Before anesthesia induction, 4.4ml(32mg） was given by a single intravenous injection, which was completed within 30 seconds
  Arms: Aprepitant Injection
Drug: Aprepitant Injection Placebo — Before anesthesia induction, 4.4ml was given by a single intravenous injection, which was completed within 30 seconds
  Arms: Aprepitant Injection Placebo

SUMMARY:
The goal of this Interventional study is to evaluate the efficacy and safety of Aprepitant Injection(QLG2174) for preventing PONV in Chinese patients.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 to 70 years, with a body mass index (BMI) of 18-30 kg/m² and body weight≥45kg.
* laparoscopic gynecologic or abdominal surgery under general anesthesia (duration≥1 hour and postoperative hospitalization ≥24 hours), with anesthesia maintained using sevoflurane and remifentanil (propofol maintenance was prohibited);
* had≥2 risk factors of PONV; expected to use postoperative opioid within 24 hours after surgery;
* American Society of Anesthesiologists (ASA) physical status class I-III.

Exclusion Criteria:

* planned intrathoracic, transplant, or central nervous system surgeries;
* diagnostic-only procedures;
* use of local/regional anesthesia (e.g., neuraxial/nerve blocks);
* postoperative intensive care unit (ICU) transfer;
* preoperative nasogastric/orogastric tube placement (from screening through 24 hours postoperatively)
* nausea, vomiting, retching, or organic disease-related emesis (e.g., intestinal obstruction) within 24 hours preoperatively; history of malignancy, epilepsy, or vestibular dysfunction;
* hypersensitivity to aprepitant;
* recent use of aprepitant/NK1 antagonists (within 2 weeks prior to randomization), antiemetics (including 5-HT3 antagonists, corticosteroids; within 1 week), strong CYP3A4 inhibitors/substrates (within 1 week), CYP3A4 inducers (within 4 weeks), or warfarin (within 2 weeks);
* clinically significant laboratory abnormalities (ALT/AST ≥2×upper limit of normal [ULN], total bilirubin ≥1.5×ULN, creatinine ≥1.5×ULN, hemoglobin ≤90 g/L)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 518 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Complete response (CR) rates over 24 hours after the end of surgery | 0-24 hours after the end of surgery
  Complete response (defined as no emetic episodes and no use of rescue therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology, Wuhan, China